CLINICAL TRIAL: NCT01891448
Title: Impact of an Intervention Using a Web-based Tool to Improve the Reporting of Randomized Controlled Trials
Brief Title: Web-based Tool to Improve Reporting of Randomized Controlled Trials
Acronym: WebCONSORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RAV008
Record Dates: First submitted 2013-05-24; First posted 2013-07-03 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Randomized Controlled Trial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- WebCONSORT tool (Experimental): This WebCONSORT tool allows authors to combine different extensions relevant to their trial and generate a list of items and a flowchart specific to their trial design and the type of intervention tested.
  Interventions: Other: WebCONSORT tool
- Modified WebCONSORT tool (Other): This tool will include the flowchart part of the WEBCONSORT tool but not the main checklist or elements relating to CONSORT extensions.
  Interventions: Other: Modified WebCONSORT tool

INTERVENTIONS:
Other: WebCONSORT tool — Authors are directed to the WebCONSORT tool. The tool allows authors to obtain a customized CONSORT checklist and flow diagram specific to their trial design (e.g., non-inferiority trial, pragmatic trial, cluster trial) and type of intervention (e.g., pharmacological or non pharmacological). The checklist items and flow diagram should then be reported in the manuscript and the completed checklist submitted to the journal along with the revision.
  Arms: WebCONSORT tool
Other: Modified WebCONSORT tool — Authors are directed to a different version of the WebCONSORT tool. This tool includes the flow diagram part of the tool but not the main checklist or elements relating to CONSORT extensions.
  Arms: Modified WebCONSORT tool

SUMMARY:
The CONSORT (Consolidated Standards of Reporting Trials) Statement aims to improve the reporting of randomized trials. If trials are not well reported it is difficult for clinicians to use best evidence to inform clinical practice and patients may not get the best care. A number of different CONSORT extensions have been developed which specify additional information needed for more complex trials. The aim of this project is to evaluate whether using a simple web-based tool (WEBCONSORT) improves the reporting of clinical trials. The tool combines different CONSORT extensions and allows authors to obtain a checklist and flow diagram which is specific to their individual trial. In this study authors of participating journals are requested, at the manuscript revision stage, to use a web-based tool to improve the reporting of their randomized trial. Authors registering to use the tool are randomized to intervention or control. In the intervention group authors are directed to the WebCONSORT tool. In the control group, authors are directed to a different version of the WebCONSORT tool which includes the flow diagram part of the tool but not the main checklist or elements relating to CONSORT extensions. The aim is that this tool should lead to improvements in the reporting of randomized trials, making it easier for clinicians to read and interpret published findings.

DETAILED DESCRIPTION:
The CONSORT (Consolidated Standards of Reporting Trials) Statement (www.consort-statement.org) is an evidence based guideline which aims to improve the reporting of randomized controlled trials. If trials are not well reported it is difficult for clinicians to use best evidence to inform clinical practice and patients may not get the best care. A number of different CONSORT extensions have been developed which specify additional information needed for more complex trials.We are conducting a multicentre randomized controlled trial to evaluate whether using a simple web-based tool (WebCONSORT) improves the completeness of reporting of clinical trials. To be eligible for inclusion in this study journals must publish reports of randomized trials and endorse the CONSORT Statement (e.g. refer to it on the journal website) but do not actively implement it (e.g. require authors to submit a completed CONSORT checklist at the time of manuscript submission. Participating journals ask authors to register their manuscript (at the revision stage of the manuscript) on the WebCONSORT website where he or she will be randomized into one of two groups (i.e. intervention and control). In the intervention group, authors will be directed to the WebCONSORT tool. The tool allows authors to combine different extensions relevant to their trial and generate a list of items and a flowchart specific to their trial design and the type of intervention tested. The checklist of items generated by the WebCONSORT tool should then be reported in the revised paper and the completed checklist and flow diagram submitted to the journal along with the revised manuscript.In the control group, authors will be directed to a different version of the WebCONSORT tool. This tool will include the flowchart part of the WEBCONSORT tool but not the main checklist or elements relating to CONSORT extensions. The primary outcome measure is the percentage of poorly reported methodological items in the submitted manuscript. Secondary outcomes include time spent on the WEBCONSORT website, rejection rate of studies, feedback from authors and compliance rate. It is anticipated that the web-based tool will lead to improvements in the reporting and transparency of trial findings, thus aiding their critical appraisal and interpretation by readers.

ELIGIBILITY:
Inclusion Criteria:

* Journals which publish reports of randomized trials and endorse the CONSORT Statement (e.g. refer to it on the journal website) but do not actively implement it (e.g. require authors to submit a completed CONSORT checklist at the time of manuscript submission).

Exclusion Criteria:

* Journals which endorse the CONSORT Statement (e.g. refer to it on the journal website) and actively implement it (e.g. require authors to submit a completed CONSORT checklist at the time of manuscript submission).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2013-03-25 (Actual); Primary Completion 2015-09-22 (Actual); Study Completion 2015-09-22 (Actual)

PRIMARY OUTCOMES:
Completeness of reporting | Following manuscript revision at 3 months
  The proportion of most poorly reported CONSORT items (initial and extensions) reported in each article.

OTHER OUTCOMES:
Rejection rate | Following manuscript revision at 3 months
  The rejection rate of articles by journal.
Compliance rate | Following manuscript revision at 3 months
  The compliance rate of the authors with submitting a checklist to the journal.
Feedback | Following manuscript revision at 3 months
  Feedback from authors on the review process after the editor's decision, and feedback from journal editors.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Ravaud, PhD, Principal Investigator — Université Paris Descartes
Locations (2):
- Université Paris Descartes, Paris, France
- University of Oxford, Oxford, United Kingdom

REFERENCES:
- [Derived] Hopewell S, Boutron I, Altman DG, Barbour G, Moher D, Montori V, Schriger D, Cook J, Gerry S, Omar O, Dutton P, Roberts C, Frangou E, Clifton L, Chiocchia V, Rombach I, Wartolowska K, Ravaud P. Impact of a web-based tool (WebCONSORT) to improve the reporting of randomised trials: results of a randomised controlled trial. BMC Med. 2016 Nov 28;14(1):199. doi: 10.1186/s12916-016-0736-x. PMID 27894295